CLINICAL TRIAL: NCT04602819
Title: Photoaging Reversing After Picosecond Laser With Diffractive Focus Lens Assessed by Cellular Resolution Optical Coherent Tomography in Asian Patient With Melasma
Brief Title: Photoaging Reversing After Picosecond Laser With DLA Assessed by Cellular Resolution OCT in Asian Patient With Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Principal Investigator, Chang Chang Cheng, Director, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH109-REC3-125
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Melasma
Keywords: basement membrane; diffractive lens array; melasma; optical coherence tomography; 755nm picosecond alexandrite laser; photoaging; vascularization; VISIA®
MeSH Terms: conditions — Melanosis; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: PicoSure 755nm picosecond alexandrite laser with diffractive lens; Device: ApolloVue® S100 Image System; Device: Cutometer® dual MPA 580; Device: VISIA®

INTERVENTIONS:
Device: PicoSure 755nm picosecond alexandrite laser with diffractive lens — Understand the role of 755nm picosecond alexandrite laser with diffractive lens of reversal of photodamage and improving the melasma by evaluation with optical coherence tomography and other noninvasive methods.
Device: ApolloVue® S100 Image System — Understand the role of 755nm picosecond alexandrite laser with diffractive lens of reversal of photodamage and improving the melasma by evaluation with optical coherence tomography.
  Other Names: 510(K) Number: K201552 (class II)
Device: Cutometer® dual MPA 580 — Understand the role of 755nm picosecond alexandrite laser with diffractive lens of reversal of photodamage and improving the melasma by evaluation with the Cutometer® dual MPA 580.
Device: VISIA® — Understand the role of 755nm picosecond alexandrite laser with diffractive lens of reversal of photodamage and improving the melasma by evaluation with the VISIA®.

SUMMARY:
Background Melasma is a commonly acquired hypermelanosis that affects facial sun exposed areas, most commonly in Asians and other darker skin type females. Recent evidence has demonstrated melasma to be a photoaging disorder. The histological findings of melasma are similar to photoaging and include solar elastosis, increased mast cells and sebaceous glands, as well as increased vascularization. Pendulous active melanocytes with weakened basal membranes, and changes in nuclear morphology and chromatin texture of adjacent basal keratinocytes also seemed to be a characteristic feature of melasma.

Objectives:

To compare the difference of photoaging features of melasma skin and normal skin by optical coherence tomography (ApolloVue® S100 Image System, a 510(K) class II medical device) and reversal of photoaing features by 755nm picosecond alexandrite laser with diffractive lens.

Methodology:

We enroll 20 adults with facial melasma. The patients received 755nm picosecond alexandrite laser with diffractive lens array over whole face at W0, W4, and W8. Evaluation with VISIA, optical coherence tomography, Cutometer MPA580 at W4, W8, W12. All the patients will be instructed with use of moisturizer, gentle cleaning, and sunscreen use.

Anticipated results and applications:

This study expects to

1. understand the role of 755nm picosecond alexandrite laser with diffractive lens of reversal of photodamage and improving the melasma by evaluation with optical coherence tomography and other noninvasive methods.
2. Set evidence based guidance for melasma treatment and set the protocol or clinical path.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written inform consent form
* Adults over the age of 20.
* Patients with melasma on their faces.

Exclusion Criteria:

* have received any cosmetic treatments, e.g. laser, pulsed light, and chemical peels within six months before participating the trial.
* Have taken oral contraceptives or received hormone therapy within one year before participating the trial.
* Has other pigmented diseases or inflammatory diseases on face.
* Are pregnant or breastfeeding.
* Has conditions with poor wound healing, keloids or photosensitivity.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of melasma | 4 weeks
  Clinical improvement of melasma after picosecond laser treatment will be assessed by both physician and patient at week 0, week 4, week 8, and week 12.
Improvement of MASI score | 4 weeks
  Improvement of melasma after picosecond laser treatment will be assessed using MASI score that will be calculated according to the image taken by VISIA at week 0, week 4, week 8, and week 12.
Improvement of hydration, TEWL, viscoelasticity, or melanin and erythema index | 4 weeks
  Improvement of melasma after picosecond laser treatment will be assessed using Cutometer® MPA 580 at week 0, week 4, week 8, and week 12.
Number of subjects with clear tissue characteristics of melasma and/or normal skin in tomograms | 4 weeks
  Number of subjects with clear tissue characteristics of tomograms will be compared to that with unclear tissue characteristics to identify the effect of the OCT on scanning melasma at study completion.

SECONDARY OUTCOMES:
Number of subjects with the distinction between melasma and normal skin in tomograms | 1 year
  Number of subjects with the distinction between melasma and normal skin in tomograms will be compared to that with no distinction to verify the specific diseases that can be distinguished from others by the OCT at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Cheng Chang, M.D., Ph. D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YJ, Chang CC, Wu YH, Huang L, Shen JW, Lu ME, Chiang HM, Lin BS. Adaptability of melanocytes post ultraviolet stimulation in patients with melasma. Lasers Surg Med. 2023 Sep;55(7):680-689. doi: 10.1002/lsm.23699. Epub 2023 Jun 27. PMID 37365922